CLINICAL TRIAL: NCT07076342
Title: Mechanistic Clinical Trial Evaluating the Role of the Metabotropic Glutamate Receptor Subtype 5 (mGluR5) in the Antidepressant Mechanism of Cognitive Behavioral Therapy for Insomnia (CBT-I)
Brief Title: The Role of mGluR5 in CBT-I
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Stony Brook University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Christine DeLorenzo, Professor of Psychiatry & Biomedical Engineering, Director (CUBIT), Stony Brook University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-00015; 1R01MH137211-01A1 (NIH)
Record Dates: First submitted 2025-07-14; First posted 2025-07-22 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Major Depressive Disorder (MDD)
Keywords: Cognitive Behavioral Therapy; CBT-I; Cognitive Behavioral Therapy & Insomnia; Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major; Sleep Initiation and Maintenance Disorders | interventions — Cognitive Behavioral Therapy; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Intervention Model Description: Prior to and following CBT-I, the investigators will quantify hippocampal mGluR5 density (with PET using [11C]ABP688) and sleep latency (with polysomnography study performed in a Sleep Lab Facility), CBT-I will be delivered through an online program, Sleep Healthy Using The Internet (SHUTi, pronounced "shut eye").
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cognitive Behavioral Therapy for Insomnia Treatment Arm (Experimental): Cognitive Behavioral Therapy for Insomnia (CBT-I) will be delivered through an online program, Sleep Healthy Using The Internet (SHUTi).
  Interventions: Behavioral: Cognitive Behavioral Therapy for Insomnia; Drug: PET Scan with [11C]ABP688

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for Insomnia — Cognitive Behavioral Therapy for Insomnia (CBT-I) will be delivered through an online program, Sleep Healthy Using The Internet Sleep Healthy Using The Internet (SHUTi)
Drug: PET Scan with [11C]ABP688 — Prior to and after completing the CBT-I protocol, participants will undergo a PET scan using tracer [11C]ABP688) to quantify hippocampal mGluR5 density.

SUMMARY:
This is mechanistic clinical trial that evaluates the role of one of the glutamate receptors (mGluR5) in cognitive behavioral therapy for insomnia (CBT-I) as a common pathway in improving sleep and depression.

DETAILED DESCRIPTION:
Cognitive behavioral therapy for insomnia (CBT-I), a treatment solely aimed at improving sleep, reduces depression with rates similar to conventional antidepressants. Although this efficacy reflects the interrelationship between sleep and depression, CBT-I's antidepressant mechanism of action is currently unknown. One potential mechanistic pathway is through the metabotropic glutamate receptor subtype 5 (mGluR5), due to its strong association with both depression and sleep. The investigators hypothesize that CBT-I's antidepressant efficacy may occur through the downregulation of mGluR5 associated with improved sleep. This study is a mechanistic clinical trial in a cohort of adults with MDD and a range of sleep latencies (time it takes to fall asleep). Prior to and following CBT-I, the investigators will quantify hippocampal mGluR5 density (with using positron emission tomography [PET] imaging) and sleep latency (with polysomnography performed in the Sleep Lab). CBT-I will be delivered through an online program, Sleep Healthy Using The Internet (SHUTi).

ELIGIBILITY:
Inclusion Criteria:

* capacity to provide informed consent,
* at least 18 years of age
* good physical health and absence of significant medical conditions,
* diagnosis of major depressive disorder (MDD) with current major depressive episode as per DSM-5 criteria
* Montgomery-Åsberg Depression Rating Scale (MADRS) score > 29 (at least moderate depression),
* uniform range of sleep latencies up to 128 minutes.

Exclusion Criteria:

* currently taking effective antidepressants,
* lifetime history of psychosis,
* drug or alcohol dependence in the last 6 months or abuse in the last 2 months
* unstable medical condition (i.e., condition not adequately stabilized for ≥ 3 months)
* nicotine use within 1 year
* currently on medication known to affect glutamate,
* sleep disorders, other than insomnia, such as sleep apnea,
* recent (within 1 year) regular night shift work (or rotating shift work) or recent (within 3 months) travel across more than one time zone, or plans for this work or travel during the study period,
* use of medication or substances that affect sleep, for example, ingestion of more > 600 mg of caffeine per day,
* PET or MRI contraindications, including pregnancy or currently breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2030-06 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Change in Sleep Latency from Baseline to 8 Weeks | Baseline and 8 Weeks
  Polysomnography: Prior to and following CBT-I, participants will spend one or two nights in the facility's Sleep Lab in order to assess sleep latency (i.e., quantity of sleep). While the participant sleeps, polysomnography, including EEG will be collected. This will be used to quantify sleep latency.
Change from Baseline of mGluR5 density in the hippocampus after 8 weeks of CBT-I Treatment | Baseline and 8 weeks
  PET Imaging: Prior to and following CBT-I, participants will receive PET imaging to allow measurement of change in mGluR5 (a protein receptor in the brain) density in the hippocampus.

CONTACTS AND LOCATIONS:
Locations (1):
- Stony Brook University: Dept of Psychiatry, Stony Brook, New York, United States